CLINICAL TRIAL: NCT00233688
Title: A Prospective, Multicenter Study of the Cordis Endovascular QUANTUM LP™ Stent Graft System for the Treatment of Abdominal Aortic Aneurysms (AAA)-FORTRON
Brief Title: Study of the Endovascular QUANTUM LP™ Stent Graft System in Abdominal Aortic Aneurysms (AAA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: H. Wayne Hutman, MD / Director, Cordis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01-4601
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): QUANTUM LP™ STENT GRAFT SYSTEM
  Interventions: Device: QUANTUM LP™ STENT GRAFT SYSTEM
- 2 (Active Comparator): Surgical intervention
  Interventions: Procedure: Open surgical repair

INTERVENTIONS:
Device: QUANTUM LP™ STENT GRAFT SYSTEM — Stent Graft System for the Treatment of Abdominal Aortic Aneurysms
  Arms: 1
Procedure: Open surgical repair — Open surgical repair
  Arms: 2

SUMMARY:
The objective of this clinical study is to assess the safety and effectiveness of the Cordis Endovascular Quantum LP™ Stent Graft System.

ELIGIBILITY:
Inclusion Criteria (Surgical Patients):

1. Non-emergent surgical candidate (aneurysm has not ruptured)
2. Patients 21 years of age or older
3. Male or infertile Female
4. Aneurysm >/=4.5 cm in diameter, or
5. Aneurysm >/= twice the normal aortic diameter directly above the aneurysm, or
6. Aneurysm >/= 4.0 cm in diameter and rapidly growing (0.5 cm in 6 months), or
7. Saccular aneurysm > 3.0 cm

Inclusion Criteria (Stent Graft Patients)

1. Patient meets all inclusion criteria for surgical candidate
2. Aneurysm starts >/= 10 mm below the most distal main renal artery and the diameter of aorta within that aortic neck segment is not variable
3. Diameter of aortic fixation zone (neck) >/= 22mm and </= 30 mm
4. Supra renal aortic diameter </= 34 mm
5. The required device coverage length >/= 13 cm extending from most distal main renal artery ostium to the distal anchoring site within the common iliac artery (or external iliac artery if planned occlusion of internal iliac artery)
6. Aortic neck angulation < 60° as estimated from CT scan images or angiogram
7. Iliac artery attachment zone diameter </= 20 mm
8. Iliac arteries with a length of >/= 10 mm of non-aneurysmal vessel located at the iliac graft attachment sites
9. Iliac arteries with adequate peripheral access to accommodate a 22 Fr catheter delivery system
10. Aortic bifurcation > 18 mm in diameter
11. Creatinine level < 2.5 mg/dl

Exclusion Criteria (Surgical and Stent Graft Patients):

1. Weight > 350 lbs. (159 Kg)
2. Mycotic, ruptured or traumatic aneurysm
3. Life expectancy < 2 years
4. MI, cerebral vascular accident or transient ischemic attack (TIA) within 6 months
5. Expected occlusion or the need for re-implantation of significant mesenteric or renal arteries originating from the AAA

Exclusion Criteria (Stent Graft Patients only)

1. Aneurysm is symptomatic or tender
2. Creatinine > 2.5 mg/dl or patient on dialysis
3. Thrombus in proximal and distal attachment area covering greater than 50% of the endoluminal surface

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2001-11; Primary Completion 2004-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To compare the aneurysm-related one-year mortality rates of the stent graft patients to open surgery patients. The purpose of having an aneurysm surgically or endovascularly repaired is to prevent death from AAA. | One year
To compare the one-year procedure-related severe adverse event rates of the stent graft patients to open surgery patients. These events exclude aneurysm-related deaths. The endpoint for this objective will be the occurrence of any serious adverse eve | One year

SECONDARY OUTCOMES:
To evaluate the occurrence of severe device-related adverse events as they relate to the cause of aneurysm exclusion failures (i.e., Type I and III endoleaks, significant AAA growth, or AAA rupture). | 30 days, 6 mo, and annually up to five years
To compare the rate and amount of blood products used in the stent graft procedure to open surgery. | At procedure

CONTACTS AND LOCATIONS:
Overall Officials: H. Wayne Hutman, MD, Study Director — Cordis US Corp.
Locations (1):
- Newark Beth Israel Medical Center, Newark, New Jersey, United States